CLINICAL TRIAL: NCT04018053
Title: A Pilot Study of 18Fluorine-Fluciclovine Positron Emission Tomography/Computed Tomography for Staging Muscle Invasive Bladder Cancer Preceding Radical Cystectomy
Brief Title: 18Fluorine-Fluciclovine PET/CT for Staging Muscle Invasive Bladder Cancer Preceding Radical Cystectomy
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Blue Earth Diagnostics (Industry)
Responsible Party: Principal Investigator, Heather A. Jacene, MD, Principal Investigator, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-208
Record Dates: First submitted 2019-07-10; First posted 2019-07-12 (Actual); Results first posted 2026-01-09 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Bladder Cancer; Urothelial Carcinoma
Keywords: Bladder cancer; urothelial carcinoma; cystectomy
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell | interventions — fluciclovine F-18; Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 18F-fluciclovine (Experimental): * 18F-fluciclovine will be administered via slow push over 10 seconds through a peripheral intravenous line
  * Immediately after the injection of the radiopharmaceutical, dynamic PET/CT images of the pelvis will be obtained for 15 minutes
  * Subsequently, PET/CT images will be obtained from the pelvis to the base of skull.
  Interventions: Drug: 18F-fluciclovine; Device: PET/CT

INTERVENTIONS:
Drug: 18F-fluciclovine — 18F-fluciclovine is a new radiotracer. This radiotracer targets amino-acid transporters, which are overexpressed in multiple cancers.
  Other Names: Axumin
Device: PET/CT — Positron emission tomography/computed tomography (PET/CT) uses small amounts of radioactive materials called radiotracers, a special camera and a computer to help evaluate organ and tissue functions.

SUMMARY:
This research study is studying a positron emission tomography (PET) agent called 18F-fluciclovine to evaluate how well 18F-fluciclovine-PET scans determine the extent of muscle invasive bladder cancer (as compared to regular CT and MRI imaging) and whether 18F-fluciclovine-PET scans can provide information about the pathologic grade of the tumor.

DETAILED DESCRIPTION:
This research study is a pilot study, which is the first-time investigators are examining this study imaging agent, 18F-fluciclovine, for use in imaging bladder cancer.

Staging of muscle invasive bladder cancer is currently done using computed tomography (CT) and/or magnetic resonance imaging (MRI). Both CT and MRI are useful to determine the extent of bladder cancer, but some studies show that up to 40% of patients with negative CT or MRI scans for disease outside the bladder are found to have disease outside the bladder (in lymph nodes near the bladder) at the time of surgery.

Given the limitations of the imaging exams currently used for staging bladder cancer, new techniques and imaging agents that can better identify metastatic lesions, especially within the pelvis, are desired and would be very useful.

18F-fluciclovine is a new radiotracer that was recently approved to evaluate lesions in recurrent prostate cancer (but not for bladder cancer). This radiotracer targets amino-acid receptors, which are overexpressed in multiple cancers. Studies have shown that 18F-fluciclovine PET/CT can visualize other types of cancers, such as breast cancer. A major advantage of 18F-fluciclovine is that it does not get into the bladder during the time of imaging. This may make it easier to see disease in the pelvis that is outside the bladder.

The purpose of this study to determine whether 18F-fluciclovine PET/CT can better stage muscle invasive bladder cancer compared to conventional CT or MRI. A secondary aim of this study is to determine whether 18F-fluciclovine PET/CT can reveal the pathologic grade of the bladder cancer, which is only determined from pathology specimens obtained at surgery.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed urothelial carcinoma of the bladder.
* Participants must have cT2-T4N0 disease at the time of the study, as defined by conventional CT or MRI imaging. Patients must have no definite evidence of locoregional or distant metastatic disease at the time of study eligibility, as defined by conventional imaging.
* Radical cystectomy must be planned for the patient after the planned 18F-fluciclovine-PET/CT.
* Patients may or may not have had prior neoadjuvant therapy prior to this study.
* Age ≥18 years. Since no dosing or adverse event data are currently available on the use of 18F-fluciclovine in participants <18 years of age, and the majority of bladder cancer occur in the adult population [42], children are excluded from this study but will be eligible for future pediatric trials.
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A)
* Ability and willingness to comply with the study procedures.
* The effects of 18F-fluciclovine on the developing human fetus are unknown. For this reason and because radiopharmaceuticals may be teratogenic, women of childbearing potential and men must agree to use adequate contraception (barrier method of birth control; abstinence) prior to study entry and for 24 hours after the PET/CT scan is completed. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Participants with other known malignancies that has required treatment in the past 3 years.
* Pregnant women are excluded from this study because 18F-fluciclovine is a radiopharmaceutical with the potential for teratogenic effects. Because of the radiation exposure to a nursing infant from 18F-fluciclovine, women who are breastfeeding are also excluded from this study.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to 18F-fluciclovine.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Contraindications for PET/CT including:

  * Severe claustrophobia
* Any past or current condition that in the opinion of the study investigators would confound the results of the study or pose additional risk to the patient by their participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2026-07-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Jacene, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: BCH - Contact the Technology & Innovation Development Office at www.childrensinnovations.org or email TIDO@childrens.harvard.edu BIDMC - Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu BWH - Contact the Partners Innovations team at http://www.partners.org/innovation DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu MGH - Contact the Partners Innovations team at http://www.partners.org/innovation

REFERENCES:
- [Background] Ng TSC, Liu M, Robertson M, Konik A, Cheng SC, Bakht MK, Harrington K, Wolanski A, Gilbert L, Preston M, Mossanen M, Beltran H, Hirsch MS, Sonpavde G, Jacene HA. A pilot study of [18F]F-fluciclovine positron emission tomography/computed tomography for staging muscle invasive bladder cancer preceding radical cystectomy. Eur J Nucl Med Mol Imaging. 2025 Sep;52(11):4092-4101. doi: 10.1007/s00259-025-07287-y. Epub 2025 Apr 21. PMID 40257614
- See also: Link to pubmed citation — https://pubmed.ncbi.nlm.nih.gov/40257614/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient consented and enrolled on 2/26/2020 until 11/2023.
Period: Overall Study
Arm/Group | 18F-fluciclovine
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: No difference between these numbers and the numbers of participants or units assigned to the arms or groups in the Participant Flow.
Groups:
- 18F-fluciclovine: Major eligibility criteria were histologically or cytologically confirmed MIBC, clinical stage T2-T4, N0 disease by CT/MRI at the time of study enrollment, and planned RC. Participants may or may not have had neoadjuvant systemic therapy before enrollment and prior to RC.
Arm/Group | 18F-fluciclovine
Number analyzed (Participants) | 16
Age, Continuous [Median (Full Range); unit: years] — Age of participant
  years | 73 [57 to 88]
Sex: Female, Male [Count of Participants; unit: Participants] — Number of participants
  Participants
    Female | 5
    Male | 11
Lymph node metastases detection with fluciclovine PET in muscle-invasive bladder cancer [Count of Participants; unit: Participants] — Fluciclovine PET and pathology agreed for 12 of 16 participants about pelvic lymph node metastases being present or absent.
  Participants | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: The Agreement Rate of Metastatic Disease Status Between 18F-fluciclovine-PET/CT and Histopathology From Radical Cystectomy
Description: Lymph nodes will be classified as positive or negative for metastatic disease on 18F-fluciclovine PET/CT and compared to pathologic stage as determined from surgery.
Time Frame: 2 years
Population: 16 patients with muscle-invasive bladder cancer who underwent radical cystectomy; 12 with prior neoadjuvant chemotherapy before radical cystectomy.
Measure: Number (95% Confidence Interval); unit: proportion of agreement scan and path
Arm/Group | 18F-fluciclovine
Number analyzed (Participants) | 16
proportion of agreement scan and path | 0.67 [0.44 to 0.83]

2. Secondary Outcome: The Amount of 18F-fluciclovine Accumulation in the Primary Bladder Tumor on PET
Description: 18F-fluciclovine SUVmax in primary bladder tumor as a measure of uptake; primary tumor stage and size at radical cystectomy
Time Frame: 2 years
Reporting Status: Not Posted

3. Secondary Outcome: Number of Participants With Suspected Distant Metastatic Disease by 18F-fluciclovine-PET/CT
Description: Visualization of distant metastases on 18F-fluciclovine-PET/CT will be binary-categorized as present/absent. We will compute sensitivity to compare 18F-fluciclovine-PET/CT with standard imaging modalities for distant metastases. The number of distant metastases will be descriptively shown by imaging modalities.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | 18F-fluciclovine
Number analyzed (Participants) | 16
participants | 0

4. Secondary Outcome: 18F-fluciclovine Uptake on PET/CT to the Presence/Absence of ASCT2 and LAT1 Amino Acid Transporters.
Description: 18F-fluciclovine SUVmax in primary bladder tumor; Presence/absence of ASCT2 and LAT1 amino acid transporter in resected primary bladder tumors
Time Frame: 2 Years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All adverse events were recorded for each participant for 24 hours after injection of the radiotracer (i.e., F18-fluciclovine)
Description: Adverse events were collected from the time of injection until 24 hours after the administration of F18-fluciclovine. Adverse events from standard of care imaging and beyond 24 hours from the injection/scan were not collected.
Arm/Group | 18F-fluciclovine
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-10): https://cdn.clinicaltrials.gov/large-docs/53/NCT04018053/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-06): https://cdn.clinicaltrials.gov/large-docs/53/NCT04018053/ICF_001.pdf